CLINICAL TRIAL: NCT01234974
Title: Phase II Study of the IGF-1 Inhibitor Pasireotide Lar in Combination With the m-TOR Inhibitor Everolimus in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: IGF-1 Inhibitor Pasireotide Lar in Combination With the m-TOR Inhibitor Everolimus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never undertaken
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Giampaolo Talamo, Associate Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSHCI 09-095
Record Dates: First submitted 2010-08-24; First posted 2010-11-04 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pasireotide; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pasireotide (Experimental): Pasireotide 60 mg day 1 every 28 days
  Interventions: Drug: Pasireotide; Drug: Everolimus

INTERVENTIONS:
Drug: Pasireotide — Given as an intramuscular injection on day 1 every 28 days, 60 mg per dose
  Other Names: Pasireotide s.c.; Pasireotide LAR; SOM230
Drug: Everolimus — given as an oral tablet every day on days 1-28, 10 mg per day
  Other Names: RAD001

SUMMARY:
Observe the safety/tolerability and effectiveness in terms of response rate and duration of response of the combination pasireotide + everolimus in the treatment of patients with relapsed/refractory multiple melanoma.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a B-cell malignancy of plasma cells. It represents the second most common hematological malignancy, with non-Hodgkin's lymphoma being the most common.In this protocol, we propose a regimen consisting of a novel combination of two agents with a promising preclinical activity, i.e., pasireotide (IGF-1 inhibitor) and everolimus (mTOR inhibitor), exploring the efficacy of this therapy in patients with MM. We propose enrollment after failure to the first two lines of FDA-approved agents, even in patients who did not have high-dose chemotherapy and SCT. In fact, overall survival after SCT has been shown to be identical when "early" SCT is compared to "late" SCT, i.e., administered at the time of relapse. This provides an important opportunity to test our novel therapeutic approach, reserving SCT for relapse. The advantage of the this strategy is that similar overall survival outcomes can be achieved with fewer patients undergoing SCT. Both everolimus and pasireotide have the potential of being clinically effective against myeloma. A phase II trial of the mTOR inhibitor temsirolimus, an analogue of everolimus, produced a response rate of 38% in relapsed/refractory multiple myeloma. The IGF-1 inhibitor pasireotide is a promising agent, because IGF has been recently found to be one of the most important growth signal molecule in myeloma cells. The combination of everolimus and pasireotide should have a synergistic antimyeloma effect because preclinical data invitro have shown that combined inhibition of mTOR inhibition and IGF-1 led to a synergistic increase of cell growth inhibition in multiple myeloma cells and might represent a potential new treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented multiple myeloma
* Multiple myeloma relapsing or refractory to at least 2 of the currently accepted therapies for multiple myeloma
* Age > 18 years
* Minimum of 4 weeks since any major surgery, radiation or 5 half life since prior systemic anticancer therapy
* ECOG performance status ≤ 2
* Anticipated life expectancy of 12 weeks or more
* Adequate bone marrow function
* Adequate liver function
* Calculated creatinine
* INR ≤ 1.5
* Fasting serum cholesterol ≤ 300 mg/dL or ≤ 7.75 mmol/L and fasting triglycerides ≤ 2.5 x ULN
* Women of childbearing potential must have a negative serum pregnancy test. Women must not be lactating. Both men and women of childbearing potential must be advised of the importance of using effective birth control during the course of the study.

Exclusion Criteria:

* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period.
* Patients should not receive immunization with attenuated live vaccines during study period or within 1 week of study entry.
* Patients with prior or concurrent malignancy
* Patients with uncontrolled diabetes mellitus
* Patients who have congestive heart failure, unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or history of acute myocardial infarction within the 6 months preceding enrollment.
* Liver disease
* Patients who have any severe and/or uncontrolled medical condition or other conditions that could affect their participation in the study.
* Female patients who are pregnant or breast feeding, adults of reproductive potential who are not using effective birth control methods.
* Male patients whose sexual partner(s) are women of child bering potential and who are not willing to use adequate contraception during the study and for 8 weeks after the end of treatment.
* Patients with a known hypersensitivity to everolimus or other rapamycin or to its excipients.
* Known hypersensitivity to somatostatin analogues or any component of the pasireotide or octreotide LAR formulations
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol
* Patients taking medication know to inhibit, induce or be a substrate to isoenzyme CYP3A
* QTcF at screening > 450 msec, history of syncope or family history of idiopathic sudden death, sustained or clinically significant cardiac arrhythmias, risk factors for Torsades de points, concomitant disease that could prolong QT intervals, use of concomitant medications know to prolong the QT interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Primary objective | 12 patients enrolled
  Initially 12 patients will be enrolled. If there are no responses among these patients with the combination pasireotide + everolimus in the treatment the study will be terminated.

SECONDARY OUTCOMES:
Secondary objective | 25 to 37 patients enrolled
  After initial 12 patients enrolled and these patients respond, an additional 25 to 27 patients will be enrolled. We will evaluate efficacy of the combination regimen based primarily on response rate. Progression free-survival and overall survival will also be recorded and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Giampaolo Talamo, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States